CLINICAL TRIAL: NCT04423393
Title: A Phase 1, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of VIR-3434
Brief Title: Study of VIR-3434 in Healthy Volunteers and Patients With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIR-3434-1002; 2019-003837-40 (EudraCT Number)
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B Virus; Chronic Hepatitis B; HBV; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- VIR-3434 (Experimental)
  Interventions: Biological: VIR-3434
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VIR-3434 — VIR-3434 given by subcutaneous injection or intravenous infusion.
  Arms: VIR-3434
Other: Placebo — Sterile normal saline (0.9% NaCl) given by subcutaneous injection or intravenous infusion.
  Arms: Placebo

SUMMARY:
This is a Phase 1 study in which healthy volunteers and participants with chronic HBV infection will receive VIR-3434 or placebo and will be assessed for safety, tolerability, pharmacokinetics (PK), and antiviral activity (only in participants with chronic HBV infection).

ELIGIBILITY:
Healthy Volunteers:

Inclusion Criteria:

* Male or female age 18 - 55
* Weight 40-125 kg

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation
* History or evidence of drug or alcohol abuse
* History of allergic reactions to monoclonal antibodies or antibody fragments
* History of anaphylaxis

CHB Patients:

Inclusion Criteria:

* Male or female age 18 - 65
* Weight 40-125 kg
* Chronic HBV infection for >/= 6 months

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the participant unsuitable for participation
* Significant fibrosis or cirrhosis
* History or evidence of drug or alcohol abuse
* History of chronic liver disease from any cause other than chronic HBV infection
* History of hepatic decompensation
* History of anaphylaxis
* History of allergic reactions to monoclonal antibodies or antibody fragments
* History of immune complex disease
* Active infection with HIV, HCV or hepatitis Delta virus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Germany (7):
  - Investigative Site, Essen
  - Investigative Site, Frankfurt
  - Investigative Site, Hanover
  - Investigative Site, Leipzig
  - Investigative Site, Mainz
  - Investigative Site, Mannheim
  - Investigative Site, Ulm
- Investigative Site, Hong Kong, Hong Kong
- New Zealand (4):
  - Investigative Site, Auckland
  - Investigative Site, Havelock North
  - Investigative Site, Newtown
  - Investigative Site, Tauranga
- Investigative Site, Bucharest, Romania
- Investigative Site, Singapore, Singapore
- South Korea (2):
  - Investigative Site, Busan
  - Investigative Site, Seoul
- United Kingdom (3):
  - Investigative Site, Birmingham
  - Investigative Site, London
  - Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vincenzetti L, Wong R, Marzi R, Guarino B, Stefanutti E, Gupta SV, Rosen LE, Belnap DM, Wang L, Chen YP, di Iulio J, Momin A, Tracy KE, Deshpande S, Errico JM, Giovannoni F, Sprugasci N, Peter A, Seu L, Cloutier D, Tay CH, Snell G, Czudnochowski N, Lempp FA, Havenar-Daughton C, Benigni F, Lanzavecchia A, Agarwal K, Yuen MF, Wedemeyer H, Gane E, Arvin A, Corti D, Schmid MA. Engineered monoclonal antibody tobevibart enhances HBsAg capture by Fc receptor-positive cells and activates HBV-specific T cells. J Hepatol. 2026 Jan;84(1):62-73. doi: 10.1016/j.jhep.2025.08.016. Epub 2025 Aug 27. PMID 40882923

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Healthy Participants 90 mg SC: Healthy participants received 90 mg VIR-3434 subcutaneous
- Part A Healthy Participants 300 mg SC: Healthy participants received 300 mg VIR-3434 subcutaneous
- Part A Healthy Participants 900 mg SC: Healthy participants received 900 mg VIR-3434 subcutaneous
- Part A Healthy Participants 900 mg IV: Healthy Participants received 900 mg VIR-3434 intravenously
- Part A: Healthy Participants 3000 mg IV: Healthy participants received 3000 mg VIR-3434 intravenously
- Part A Healthy Participants Placebo: Healthy participants received placebo subcutaneously or intravenously
- Part B: HBV Participants 6 mg SC: HBV Participants on NRTI therapy with HBsAg <3000 IU/mL received 6 mg VIR-3434 subcutaneous
- Part B: HBV Participants 18 mg SC: HBV Participants on NRTI therapy with HBsAg <3000 IU/mL received 18 mg VIR-3434 subcutaneous
- Part B: HBV Participants 75 mg SC: HBV Participants on NRTI Therapy with HBsAg <3000 IU/mL received 75 mg VIR-3434 subcutaneous
- Part B: HBV Participants 300 mg SC: HBV Participants on NRTI Therapy with HBsAg <3000 IU/mL received 300 mg VIR-3434 subcutaneous
- Part B: HBV Participants Placebo: HBV Participants on NRTI Therapy with HBsAg <3000 IU/mL received placebo subcutaneous
- Part C: HBV Participants 18 mg SC: HBV Participants on NRTI therapy with HBsAg >/= 3000 IU/mL received 18 mg VIR-3434 subcutaneous
- Part C: HBV Participants 75 mg SC: HBV Participants on NRTI Therapy with HBsAg >/= 3000 IU/mL received 75 mg VIR-3434 subcutaneous
- Part C: HBV Participants 300 mg SC: HBV Participants on NRTI Therapy with HBsAg >/= 3000 IU/mL received 300 mg VIR-3434 subcutaneous
- Part C: HBV Participants Placebo: HBV Participants on NRTI Therapy with HBsAg >/= 3000 IU/mL received placebo subcutaneous
- Part D: HBV Participants 75 mg SC: HBV Participants not on NRTI therapy with HBV DNA >/= 1000 and any HBsAg level received 75 mg VIR-3434 subcutaneous
- Part D: HBV Participants 300 mg SC: HBV Participants not on NRTI Therapy with HBV DNA >/= 1000 and any HBsAg level received 300 mg VIR-3434 subcutaneous
- Part D: HBV Participants Placebo: HBV Participants not on NRTI Therapy with HBV DNA >/= 1000 IU/mL and any HBsAg level received placebo subcutaneous
Period: Overall Study
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part A Healthy Participants Placebo | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part B: HBV Participants Placebo | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part C: HBV Participants Placebo | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC | Part D: HBV Participants Placebo
Started | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4
Entered Extended Follow Up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 5 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 4 | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part A Healthy Participants Placebo | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part B: HBV Participants Placebo | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part C: HBV Participants Placebo | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC | Part D: HBV Participants Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (11.94) | 27.7 (7.92) | 31.5 (9.77) | 24.8 (4.58) | 29.3 (12.99) | 30.3 (10.77) | 56.3 (5.72) | 49.0 (6.93) | 50.8 (8.35) | 50.0 (8.81) | 51.6 (6.35) | 44.5 (10.82) | 38.2 (8.33) | 38.8 (8.95) | 44.0 (8.53) | 42.7 (7.71) | 38.0 (6.16) | 37.3 (8.54) | 39.6 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 5 | 4 | 6 | 0 | 0 | 2 | 1 | 1 | 3 | 2 | 2 | 3 | 4 | 3 | 2 | 49
  Male | 2 | 3 | 2 | 1 | 2 | 5 | 6 | 6 | 4 | 5 | 7 | 3 | 4 | 4 | 3 | 2 | 3 | 2 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 5 | 6 | 4 | 5 | 6 | 9 | 5 | 3 | 5 | 6 | 6 | 6 | 5 | 5 | 5 | 6 | 6 | 4 | 97
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 4 | 6 | 5 | 0 | 0 | 3 | 5 | 2 | 0 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 6
  White | 3 | 3 | 3 | 4 | 2 | 7 | 3 | 3 | 2 | 1 | 1 | 1 | 5 | 6 | 2 | 0 | 3 | 2 | 51
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 3 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 14
Baseline HbsAg (IU/mL) [Mean (Standard Deviation); unit: log 10 IU/mL] — Population: HbsAg levels would not be seen in Healthy Participants, therefore 0 participants were analyzed in Part A.
  log 10 IU/mL
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 72
    (all) |  |  |  |  |  |  | 1.94 (0.617) | 2.78 (0.711) | 2.55 (0.693) | 2.59 (1.150) | 2.24 (0.638) | 3.34 (0.455) | 4.12 (0.353) | 3.71 (0.375) | 3.18 (1.652) | 3.79 (0.729) | 4.29 (0.305) | 4.15 (0.496) | 3.17 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Treatment-emergent period, which is up to Week 24 in part A, and up to Week 8 in part B/C/D
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part A Healthy Participants Placebo | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part B: HBV Participants Placebo | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part C: HBV Participants Placebo | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC | Part D: HBV Participants Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4
Participants | 5 | 4 | 5 | 4 | 3 | 6 | 2 | 4 | 3 | 3 | 2 | 2 | 4 | 5 | 4 | 2 | 6 | 3

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Time Frame: Up to 280 days post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part A Healthy Participants Placebo | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part B: HBV Participants Placebo | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part C: HBV Participants Placebo | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC | Part D: HBV Participants Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 11 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4
Participants
  ALT Grade 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0
  ALT Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Grade 1 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
  AST Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Bilirubin Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Cmax
Description: VIR-3434 Maximum Concentration in Serum
Time Frame: Parts B-D: pre-dose and 1, 4, 6, 24 hours, 3, 7, 10, 14, 28, 56, 84, 112, 168, 224, 280 days post-dose
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Parts B-D: ng/mL
Arm/Group | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 3 | 3 | 6 | 4 | 5
Parts B-D: ng/mL | 352 (27.0) | 456 (152.8) | 5460 (36.5) | 19700 (56.9) | 835 (NA) — In the 18 mg cohort in Part C, 2 participants among the 3 who had quantifiable PK concentrations only had 2 non-BQL values, so PK parameters were excluded from summary statistics. CV% was only reported when n ≥ 3, so indicated as NA in this case. | 4750 (46.9) | 26100 (21.8) | 6000 (16.8) | 10800 (61.4)

4. Secondary Outcome: Tmax
Description: VIR-3434 time of Cmax in Serum
Time Frame: Part A: pre-dose and 1, 4, 6, 24 hours, 3, 7, 14, 28, 56, 84, 126, 168 days post-dose; Parts B-D: pre-dose and 1, 4, 6, 24 hours, 3, 7, 10, 14, 28, 56, 84, 112, 168, 224, 280 days post-dose
Population: Participants with BQL at all time points were excluded from the PK analysis, hence for different n in the cohorts. CV was only calculated if the PK parameter was estimated in at least 3 subjects
Measure: Median (Full Range); unit: day
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 3 | 3 | 6 | 4 | 5
day | 7.00 [3.00 to 7.01] | 7 [3 to 7.00] | 3 [3.00 to 7.00] | .0833 [0.0417 to 0.292] | .0833 [0.0417 to 0.0847] | 6.90 [1.01 to 7.00] | 2.92 [1.00 to 6.88] | 5.44 [2.83 to 7.03] | 2.96 [2.11 to 6.97] | 3.98 [3.98 to 3.98] | 3.00 [2.95 to 3.94] | 2.99 [2.86 to 6.97] | 4.08 [0.0417 to 8.11] | 2.99 [2.91 to 3.15]

5. Secondary Outcome: AUClast
Description: VIR-3434 under the curve from time 0 to last measurable Time
Time Frame: Parts B-D: pre-dose and 1, 4, 6, 24 hours, 3, 7, 10, 14, 28, 56, 84, 112, 168, 224, 280 days post-dose
Population: Participants with BQL at all time points were excluded from the PK analysis, hence for different n in the cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Parts B-D: day*ng/mL
Arm/Group | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 3 | 3 | 6 | 4 | 5
Parts B-D: day*ng/mL | 3130 (67.5) | 4150 (270.0) | 106000 (72.3) | 381000 (94.2) | 9540 (NA) — In the 18 mg cohort in Part C, 2 participants among the 3 who had quantifiable PK concentrations only had 2 non-BQL values, so PK parameters were excluded from summary statistics. CV% was only reported when n ≥ 3, so indicated as NA in this case. | 39000 (133.0) | 181,000 (964.4) | 9,270 (1,139.9) | 54,300 (122.7)

6. Secondary Outcome: t1/2
Description: VIR-3434 apparent Elimination Half-life (t1/2) in serum
Time Frame: as for outcome 4
Population: PK Anal;ysis Set
Measure: Median (Full Range); unit: day
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 3 | 3 | 6 | 4 | 5
day | 28.5 [27.0 to 30.3] | 24.3 [23.2 to 26.6] | 25.2 [21.6 to 28.7] | 24.0 [20.7 to 25.7] | 20.7 [19.3 to 22.7] | 3.57 [2.33 to 4.81] | 6.34 [6.34 to 6.34] | 7.94 [3.54 to 17.2] | 13.6 [5.96 to 16.0] | 3.82 [3.82 to 3.82] | 4.25 [2.48 to 6.02] | 8.36 [4.16 to 11.8] | 3.17 [3.17 to 3.17] | 1.99 [1.99 to 1.99]

7. Secondary Outcome: Vz/F
Description: VIR-3434 Volume of Distribution (SC only)
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 3 | 3 | 6 | 4 | 5
mL | 12200 (15.2) | 10900 (27.3) | 10600 (27.7) | 9420 (12.9) | 4540 (NA) — the SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA. | 7410 (21.5) | 9830 (54.2) | 10300 (NA) — the SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA. | 6710 (27.4) | 7330 (22.5) | 5000 (NA) — the SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA. | 4880 (NA) — the SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA.

8. Secondary Outcome: Vz
Description: VIR-3434 Volume of Distribution (IV only)
Time Frame: Part A: pre-dose and 1, 4, 6, 24 hours, 3, 7, 14, 28, 56, 84, 126, 168 days post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV
Number analyzed (Participants) | 6 | 6
mL | 7620 (26.3) | 7290 (24.6)

9. Secondary Outcome: CL/F
Description: VIR-3434 Apparent serum clearance (SC only)
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 3 | 3 | 6 | 4 | 5
mL/day | 295 (16.0) | 308 (22.7) | 292 (19.7) | 1950 (71.2) | 496 (NA) — The SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA. | 697 (71.6) | 653 (85.6) | 1860 (NA) — The SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA. | 1200 (111.2) | 670 (32.8) | 1090 (NA) — The SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA. | 1700 (NA) — The SAP specified that if span of < 2 half-lives or (adjusted) r2 < 0.80 or %AUCexp >20%, all elimination related parameters including Vz/F and CL/F were excluded from summary statistics. And since n<3, %CV was NA.

10. Secondary Outcome: CL
Description: VIR-3434 Apparent serum clearance (IV only)
Time Frame: Part A: pre-dose and 1, 4, 6, 24 hours, 3, 7, 14, 28, 56, 84, 126, 168 days post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV
Number analyzed (Participants) | 6 | 6
mL/day | 244 (19.6) | 1950 (71.2)

11. Secondary Outcome: Number of Participants With ADA to VIR-3434
Description: Evaluate the immunogenicity of VIR-3434
Time Frame: Part A: Up to 168 days post-dose. Parts B-D: Up to 280 days post-dose
Population: Immunogenicity Analysis Set
Measure: Number; unit: Participants
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 4 | 1

12. Secondary Outcome: Maximum Reduction of Serum HBsAg From Baseline (Day 1 Predose)
Description: HBsAg reductions at nadir and Week 4
Time Frame: Parts B-D: pre-dose and 1, 3, 7, 10, 14, 28, 56, 84, 112, 168, 224, 280 days post-dose
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part B: HBV Participants Placebo | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part C: HBV Participants Placebo | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC | Part D: HBV Participants Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4
IU/mL
  Nadir | -1.30 (0.152) | -1.27 (0.666) | -1.96 (0.436) | -2.24 (0.353) | -0.04 (0.039) | -1.05 (0.598) | -1.28 (0.749) | -2.17 (0.252) | -0.06 (0.092) | -1.77 (0.931) | -1.83 (0.219) | -0.09 (0.039)
  Week 4 | -0.61 (0.400) | -0.38 (0.503) | -1.51 (0.245) | -1.69 (0.766) | 0.02 (0.039) | -0.30 (0.382) | -0.16 (0.175) | -1.43 (0.711) | -0.01 (0.129) | -0.48 (0.608) | -0.37 (0.368) | -0.00 (0.016)

13. Secondary Outcome: Part D Only: Maximum Change of HBV DNA From Baseline (Day 1 Predose)
Description: HBV DNA reductions at nadir and Week 4
Time Frame: Parts B-D: pre-dose and 1, 3, 7, 10, 14, 28, 56, 84, 112, 168, 224, 280 days post-dose Parts B-D: pre-dose and 1, 3, 7, 10, 14, 28, 56, 84, 112, 168, 224, 280 days post-dose
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC | Part D: HBV Participants Placebo
Number analyzed (Participants) | 6 | 6 | 4
IU/mL
  Nadir | -1.44 (0.998) | -2.07 (1.007) | -0.12 (0.06)
  Week 4 | -0.70 (0.917) | -0.61 (1.195) | 0.06 (0.472)

14. Secondary Outcome: Titers (if Applicable) of ADA to VIR-3434
Description: Evaluate the immunogenicity of VIR-3434
Time Frame: Part A: Up to 168 days post-dose. Parts B-D: Up to 280 days post-dose
Population: Immunogenicity Analysis Set
Measure: Median (Full Range); unit: Median Titer
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Median Titer | 0 [0 to 0] | 20 [20 to 40] | 160 [160 to 160] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 40 [40 to 40] | 80 [40 to 160] | 240 [20 to 1280] | 120 [80 to 160] | 80 [80 to 80] | 20 [19 to 40] | 40 [20 to 2560] | 20 [20 to 320]

15. Secondary Outcome: Cmax
Description: VIR-3434 Maximum Concentration in Serum
Time Frame: Part A: pre-dose and 1, 4, 6, 24 hours, 3, 7, 14, 28, 56, 84, 126, 168 days post-dose
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Part A: μg/mL
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Part A: μg/mL | 9.46 (27.4) | 32.1 (18.0) | 105 (23.7) | 363 (32.6) | 1060 (20.00)

16. Secondary Outcome: AUClast
Description: VIR-3434 under the curve from time 0 to last measurable Time
Time Frame: Part A: pre-dose and 1, 4, 6, 24 hours, 3, 7, 14, 28, 56, 84, 126, 168 days post-dose
Population: Participants with BQL at all time points were excluded from the PK analysis, hence for different n in the cohorts. AUClast was only calculated if the PK parameter was estimated in at least 3 subjects
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Part A: day*µg/mL
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Part A: day*µg/mL | 302 (16.0) | 964 (22.6) | 3060 (19.8) | 4010 (28.5) | 12300 (19.7)

ADVERSE EVENTS:
Time Frame: Treatment-emergent period, which is up to Week 24 in part A, and up to Week 8 in part B/C/D
Arm/Group | Part A: Healthy Participants 90 mg SC | Part A Healthy Participants 300 mg SC | Part A Healthy Participants 900 mg SC | Part A Healthy Participants 900 mg IV | Part A: Healthy Participants 3000 mg IV | Part A Healthy Participants Placebo | Part B: HBV Participants 6 mg SC | Part B: HBV Participants 18 mg SC | Part B: HBV Participants 75 mg SC | Part B: HBV Participants 300 mg SC | Part B: HBV Participants Placebo | Part C: HBV Participants 18 mg SC | Part C: HBV Participants 75 mg SC | Part C: HBV Participants 300 mg SC | Part C: HBV Participants Placebo | Part D: HBV Participants 75 mg SC | Part D: HBV Participants 300 mg SC | Part D: HBV Participants Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/11 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/11 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 5/6 | 4/6 | 3/6 | 6/11 | 0/6 | 1/6 | 2/6 | 3/6 | 2/8 | 2/6 | 4/6 | 5/6 | 4/6 | 2/6 | 6/6 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Healthy Participants 90 mg SC (N=6) | Part A Healthy Participants 300 mg SC (N=6) | Part A Healthy Participants 900 mg SC (N=6) | Part A Healthy Participants 900 mg IV (N=6) | Part A: Healthy Participants 3000 mg IV (N=6) | Part A Healthy Participants Placebo (N=11) | Part B: HBV Participants 6 mg SC (N=6) | Part B: HBV Participants 18 mg SC (N=6) | Part B: HBV Participants 75 mg SC (N=6) | Part B: HBV Participants 300 mg SC (N=6) | Part B: HBV Participants Placebo (N=8) | Part C: HBV Participants 18 mg SC (N=6) | Part C: HBV Participants 75 mg SC (N=6) | Part C: HBV Participants 300 mg SC (N=6) | Part C: HBV Participants Placebo (N=6) | Part D: HBV Participants 75 mg SC (N=6) | Part D: HBV Participants 300 mg SC (N=6) | Part D: HBV Participants Placebo (N=4)
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Healthy Participants 90 mg SC (N=6) | Part A Healthy Participants 300 mg SC (N=6) | Part A Healthy Participants 900 mg SC (N=6) | Part A Healthy Participants 900 mg IV (N=6) | Part A: Healthy Participants 3000 mg IV (N=6) | Part A Healthy Participants Placebo (N=11) | Part B: HBV Participants 6 mg SC (N=6) | Part B: HBV Participants 18 mg SC (N=6) | Part B: HBV Participants 75 mg SC (N=6) | Part B: HBV Participants 300 mg SC (N=6) | Part B: HBV Participants Placebo (N=8) | Part C: HBV Participants 18 mg SC (N=6) | Part C: HBV Participants 75 mg SC (N=6) | Part C: HBV Participants 300 mg SC (N=6) | Part C: HBV Participants Placebo (N=6) | Part D: HBV Participants 75 mg SC (N=6) | Part D: HBV Participants 300 mg SC (N=6) | Part D: HBV Participants Placebo (N=4)
Headache (Nervous system disorders) | 2 | 3 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 4 | 0 | 1 | 3 | 1
Injection site erythema (General disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Leukopenia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Neutropenia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may discuss or publish results after:

* the study results in their entirety have been publicly disclosed by or with the consent of the Sponsor OR study has been completed at all investigative sites for at least 18 months.
* provision of publication up to 60 days before planned submission to allow Sponsor to remove confidential information or identify Sponsor intellectual property

Publication may be delayed as applicable, up to 120 days for Sponsor to file patent application(s)

DOCUMENTS (2):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04423393/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT04423393/SAP_001.pdf